CLINICAL TRIAL: NCT04313283
Title: Addressing Racial Disparities in Autism Diagnosis and Treatment: Translating Peer-to-Peer Support Into a Clinical Setting
Brief Title: Translating Peer-to-Peer Support Into a Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Sarah Dababnah, Associate Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00090447; 1UL1TR003098 (NIH)
Record Dates: First submitted 2020-03-15; First posted 2020-03-18 (Actual); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Development Delay; Neurodevelopmental Disorders; Autism
Keywords: Developmental delays; Parenting; Autism
MeSH Terms: conditions — Learning Disabilities; Neurodevelopmental Disorders; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parents Taking Action (Experimental): A peer-led intervention, Parents Taking Action is the psychoeducational and child behavior management intervention led by trained Parent Leaders for 12 weeks.
  Interventions: Behavioral: Parents Taking Action

INTERVENTIONS:
Behavioral: Parents Taking Action — A peer-led intervention, Parents Taking Action is the psychoeducational and child behavior management intervention led by trained Parent Leaders.

SUMMARY:
There is not a lot of research focusing on Black and African American families raising young children with developmental delays. While the investigators know that early intervention helps children and their families, Black children with developmental delays are less likely to access such services. The causes for these racial disparities are largely unknown. Researchers have recommended caregiver support programming while on waitlists to improve caregiver-provider interactions and caregiver knowledge of the diagnostic process and developmental delays. Once a child is referred to a clinic for developmental concerns, long appointment waitlists contribute to further delays in timely diagnosis and treatment, as well as parental distress. Support programs for waitlisted families can begin to address these challenges. In this study, the investigators will examine a program called Parents Taking Action with families on a waitlist for a specialty developmental evaluation. The investigators will study if the program is feasible in this setting, if participants like the program, and if child and parent outcomes improve after participants have completed the program.

DETAILED DESCRIPTION:
Partners at the University of Maryland Baltimore (UMB) School of Medicine (SOM), School of Social Work (SSW), and community collaborators will pilot an intervention focused on Black and African-American children with Autism Spectrum Disorder (hereafter, autism) and other developmental delays. The research fills several gaps in the academic literature. First, there is a dearth of intervention research focusing on Black families raising young children with autism. Early intervention significantly improves child and family outcomes across childhood and into adulthood. Yet, Black children with autism are less likely to access such services. Even when controlling for socioeconomic status, racial disparities in autism and developmental disability diagnoses and services persist. The causes for these socioeconomic and racial disparities are largely unknown. Researchers have recommended caregiver support programming while on waitlists to improve caregiver-provider interactions and caregiver knowledge of the diagnostic process; yet, such interventions have not been described in the literature.

SSW researchers led a community-based trial to adapt a peer-led intervention, Parents Taking Action, for low-income Black families raising children with autism in Baltimore. The psychoeducational and child behavior management intervention, led by trained Parent Leaders, is unique in that it considers families' cultural and socioeconomic characteristics. Our social work team worked closely with our community advisory board to make cultural adaptations to the manual for use in Baltimore with a majority Black population. Our social work team has since further adapted the program to deliver content in two six-week modules (12 weeks total).

Despite the social work team's efforts to understand and address racial autism disparities, a wholly community-based model has limitations. Once a child is referred to a clinic for developmental concerns, long appointment waitlists contribute to further delays in timely diagnosis and treatment, as well as parental distress. Wait times also contribute to appointment absenteeism, which further delays timely access to care. A study suggested support programs for waitlisted families can begin to address these challenges. In total, these studies have suggested an integrated community-clinical model can provide critical supports to children and their families while on a waitlist and strengthen connections between families and clinical providers. Thus, this project will test the feasibility, acceptability, and short-term outcomes of a peer-led program, Parents Taking Action with a clinical sample.

ELIGIBILITY:
Inclusion Criteria:

* Parent or other primary caregiver of a child age eight years or younger on University of Maryland Baltimore, Developmental-Behavioral waiting list for autism or developmental concerns
* Identify self or child as Black or African American.

Exclusion Criteria:

* Parent or other primary caregiver is younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magana S, Lopez K, Salkas K, Iland E, Morales MA, Garcia Torres M, Zeng W, Machalicek W. A Randomized Waitlist-Control Group Study of a Culturally Tailored Parent Education Intervention for Latino Parents of Children with ASD. J Autism Dev Disord. 2020 Jan;50(1):250-262. doi: 10.1007/s10803-019-04252-1. PMID 31606887
- [Background] Kuhn JL, Vanegas SB, Salgado R, Borjas SK, Magana S, Smith DaWalt L. The Cultural Adaptation of a Transition Program for Latino Families of Youth with Autism Spectrum Disorder. Fam Process. 2020 Jun;59(2):477-491. doi: 10.1111/famp.12439. Epub 2019 Mar 7. PMID 30844083
- [Background] Shaia WE, Nichols HM, Dababnah S, Campion K, Garbarino N. Brief Report: Participation of Black and African-American Families in Autism Research. J Autism Dev Disord. 2020 May;50(5):1841-1846. doi: 10.1007/s10803-019-03926-0. PMID 30805765
- [Background] Dababnah S, Shaia WE, Campion K, Nichols HM. "We Had to Keep Pushing": Caregivers' Perspectives on Autism Screening and Referral Practices of Black Children in Primary Care. Intellect Dev Disabil. 2018 Oct;56(5):321-336. doi: 10.1352/1934-9556-56.5.321. PMID 30273522
- [Background] Koegel LK, Koegel RL, Ashbaugh K, Bradshaw J. The importance of early identification and intervention for children with or at risk for autism spectrum disorders. Int J Speech Lang Pathol. 2014 Feb;16(1):50-6. doi: 10.3109/17549507.2013.861511. Epub 2013 Dec 11. PMID 24328352
- [Background] Feinberg E, Silverstein M, Donahue S, Bliss R. The impact of race on participation in part C early intervention services. J Dev Behav Pediatr. 2011 May;32(4):284-91. doi: 10.1097/DBP.0b013e3182142fbd. PMID 21389865
- [Background] Nguyen CT, Krakowiak P, Hansen R, Hertz-Picciotto I, Angkustsiri K. Sociodemographic Disparities in Intervention Service Utilization in Families of Children with Autism Spectrum Disorder. J Autism Dev Disord. 2016 Dec;46(12):3729-3738. doi: 10.1007/s10803-016-2913-3. PMID 27639855
- [Background] Mandell DS, Ittenbach RF, Levy SE, Pinto-Martin JA. Disparities in diagnoses received prior to a diagnosis of autism spectrum disorder. J Autism Dev Disord. 2007 Oct;37(9):1795-802. doi: 10.1007/s10803-006-0314-8. Epub 2006 Dec 8. PMID 17160456
- [Background] Denman K, Smart C, Dallos R, Levett P. How Families Make Sense of Their Child's Behaviour When on an Autism Assessment and Diagnosis Waiting List. J Autism Dev Disord. 2016 Nov;46(11):3408-3423. doi: 10.1007/s10803-016-2873-7. PMID 27480420
- [Background] Kalb LG, Freedman B, Foster C, Menon D, Landa R, Kishfy L, Law P. Determinants of appointment absenteeism at an outpatient pediatric autism clinic. J Dev Behav Pediatr. 2012 Nov-Dec;33(9):685-97. doi: 10.1097/DBP.0b013e31826c66ef. PMID 23095496
- [Background] Connolly M, Gersch I. A support group for parents of children on a waiting list for an assessment for autism spectrum disorder. Educational Psychology in Practice. 2013; 29(3): 293-308.
- [Derived] Dababnah S, Reyes C, Kim I, Badawi DG, Chung Y, Shaia WE. Pilot Trial of a Peer-to-Peer Psychoeducational Intervention for Parents of Black Children Awaiting a Developmental Evaluation. J Dev Behav Pediatr. 2023 Jun-Jul 01;44(5):e370-e378. doi: 10.1097/DBP.0000000000001182. Epub 2023 Apr 26. PMID 37099652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited participants whose child was waitlisted for an autism or developmental evaluation. 36 participants consented to participate in the single-arm study, but 17 of them did not receive the intervention because they did not complete baseline measures (n=12) or did not begin the intervention (n=5). Thus, 19 people began the intervention. Of these, 15 completed the intervention and all data points; the remaining 4 only completed part of the intervention and did not complete all data points.
Period: Overall Study
Arm/Group | Parents Taking Action
Started | 19
Completed | 15
Not Completed | 4
Not completed — did not complete intervention | 4

BASELINE CHARACTERISTICS:
Population: 19 people began the intervention; however, only 15 completed the intervention. The results here are based on 15 participants.
Arm/Group | Parents Taking Action
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Employment Status [Count of Participants; unit: Participants]
  Employed full-time | 5
  Employed part-time | 4
  Self-employed | 4
  Unemployed | 2
Marital Status [Count of Participants; unit: Participants]
  Never married | 8
  Married | 5
  Divorced | 1
  Other | 1
Education Level [Count of Participants; unit: Participants]
  High school graduate | 9
  College graduate | 3
  Graduate/professional school | 3
Annual Household Income (USD) [Count of Participants; unit: Participants]
  <$10,000 | 5
  $10,000 - $29,999 | 3
  $30,000 - $49,999 | 3
  $50,000 - $69,999 | 1
  ≥$70,000 | 1
  Don't know/not sure | 2

OUTCOME MEASURES:

1. Primary Outcome: Parenting Stress
Description: Autism Parenting Stress Index (APSI): This measure includes 13 items that assess core autism symptoms, comorbid behaviors, and comorbid physical behaviors. Each item is based on a 5-point rating scale with descriptors for 0, 1, 2, 3, and 5. Possible range is 0-65. Higher scores indicate more parenting stress.
Time Frame: Pre-intervention and post-intervention at 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents Taking Action
Number analyzed (Participants) | 15
score on a scale
  Pre-intervention | 14.4 (11.4)
  Post-intervention | 12.2 (8.52)

2. Secondary Outcome: Depression
Description: Center for Epidemiological Studies-Depression (CES-D)- This measure contains 20 items assess 4 separate factors: depressive affect, somatic symptoms, positive affect, and interpersonal relations. Each item is based on a 4-point rating scale with descriptors for 0, 1, 2, and 3. Possible range is 0-60. A score of 16 points or more considered depressed.
Time Frame: Pre-intervention and post-intervention at 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents Taking Action
Number analyzed (Participants) | 15
score on a scale
  Pre-intervention | 15.2 (9.7)
  Post-intervention | 10.6 (8.35)

3. Secondary Outcome: Family Functioning
Description: Family Outcomes Survey-Revised (FOS-R): This measure was developed to provide child and family outcomes for evaluation the effectiveness of early intervention program. This measure includes 24 items assessing five outcomes (1) family needs/strengths (4 items); (2) advocacy (5 items); (3) child learning support (4 items); (4) social support (5 items); and (5) community access (6 items). Each item is based on a 5-point rating scale with descriptors for 1, 2, 3, 4, and 5. Possible range is 24-120. Higher scores indicate better family functioning.
Time Frame: Pre-intervention and post-intervention at 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents Taking Action
Number analyzed (Participants) | 15
score on a scale
  Pre-intervention | 85.5 (12.3)
  Post-intervention | 99.7 (14.4)

4. Secondary Outcome: Fidelity
Description: Procedural Fidelity Checklist Self-Assessment for Promotora Home Visits: This measurement was developed to evaluate Parent Leaders' fidelity on the program delivery. This measure includes 16 items the Parent Leader completes after every program session. Each item is based on two responses: (1) I did this; (2) I did not this. Possible range is 0-100. Higher scores indicate less fidelity.
Time Frame: Weekly through intervention (12 weeks total)
Population: Parent Leaders report fidelity 0-100 on each session they have with intervention participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: intervention sessions
Arm/Group | Parents Taking Action
Number analyzed (Participants) | 15
Number analyzed (intervention sessions) | 183
score on a scale | 98 (.04)

5. Secondary Outcome: Child Behavior
Description: Nisonger Child Behavior Rating Form (NCBRF)- This measure includes 76 item in two sections, reported separately: positive social behavior and problem behavior. Each item is based on a 4-point rating scale with descriptors for 0, 1, 2, and 3.
  Section 1 (positive social behavior) contains 10 items and scores range from 0-30. Higher scores indicate more positive social behavior.
  Section 2 (problem behavior) contains 66 items and scores range from 0-198. Higher scores indicate more child behavior problems.
Time Frame: Pre-intervention and post-intervention at 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents Taking Action
Number analyzed (Participants) | 15
score on a scale
  Pre-intervention (positive social behavior total score) | 11.0 (4.4)
  Post-intervention (positive social behavior total score) | 12.1 (5.5)
  Pre-intervention (problem behavior total score) | 45.3 (32.6)
  Post-intervention (problem behavior total score) | 37.5 (19.7)

ADVERSE EVENTS:
Time Frame: We collected data on all participants while they were enrolled in the study, which lasted through completion of baseline data until post-intervention data collection (approximately 12 weeks). This single-arm was minimal risk and only involved participants engaging in a psychoeducational parenting program. In order to reduce risks and promote participant safety, we developed a Safety Plan for any emergencies or distress, as well as a Resource List for any parents seeking additional support.
Description: In the event a participant experienced emotional distress related to completing the questionnaires, the participant was asked to report the reaction to research staff. We anticipated the reactions were likely be rare, given the measures were widely utilized in clinical and research settings. However, in the event they occurred, the study team was prepared to address them on a case-by-case basis (e.g., referral to psychological services).
Arm/Group | Parents Taking Action
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT04313283/Prot_SAP_000.pdf